CLINICAL TRIAL: NCT04280796
Title: Mechanisms of Emotional-motivational Pain Processing in Health and Disease
Brief Title: Changes in Affective Pain Processing in Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: susanne becker (Other)
Collaborators: SNSF (Unknown)
Responsible Party: Sponsor-Investigator, susanne becker, Head of Research Group, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PR00P1_179697/1
Record Dates: First submitted 2020-01-15; First posted 2020-02-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pain, Acute; Pain, Chronic; Low Back Pain
Keywords: acute pain; chronic pain; low back pain; hedonic shift; emotional-motivation components of pain; sensory-discriminative components of pain; operant conditioning; metacognition
MeSH Terms: conditions — Acute Pain; Chronic Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Study comprises an intervention that is neither a therapeutic or transplant product nor a transplant. Study involves minimal risks for participants. Used methods are within the range of standard methods frequently used in pain research. All participants will perform 2 psychophysical tasks to assess sensory-discriminative & emotional-motivational pain responses independently from each other.
  Substudy1: An operant learning paradigm will be implemented to dissociate these responses, increasing the sensory-discriminative compared to emotional-motivational pain responses by contingent monetary reinforcement & vice versa. Substudy2: Responses of chronic pain patients will be compared to those of healthy participants to characterize possible alterations. Operant learning will be operationalized to decrease emotional-motivational pain responses, which are assumed to be increased in patients. Substudy3: Participants will perform a psychophysical task to assess metacognition in pain perception.
Who Masked: Participant
Masking Description: participants are not fully instructed about the purpose before and during the test but will be debriefed after testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Substudy 1 (Experimental): All participants will perform two psychophysical tasks to assess sensory-discriminative and emotional-motivational pain responses independently from each other. No arms will perform. In addition, in Substudy 1 an operant learning paradigm will be implemented to dissociate these responses, increasing the sensory-discriminative pain responses compared to emotional-motivational pain responses by contingent monetary reinforcement and vice versa.
  Primary objectives:
  1. To develop psychophysical methods that allow the independent assessment of sensory-discriminative and emotional-motivational pain responses and
  2. to show that emotional-motivational and sensory-discriminative pain components can be dissociated
  Secondary objective:
  To assess whether fear of pain, fear-avoidance beliefs, pain catastrophizing, and sensation seeking as personality traits can explain variations in how strongly sensory-discriminative and emotional-motivational pain responses can be dissociated
  Interventions: Behavioral: psychophysical tasks
- Substudy 2 (Experimental): All participants will perform two psychophysical tasks to assess sensory-discriminative and emotional-motivational pain responses independently from each other. No arms will perform. In addition, in Substudy 2, responses of chronic pain patients will be compared to those of healthy participants to characterize possible alterations in the patients and operant learning will be operationalized to decrease emotional-motivational pain responses, which are assumed to be already increased in the patients.
  Primary objective:
  To demonstrate that in chronic pain patients, emotional-motivational pain responses are increased relative to sensory-discriminative pain responses
  Secondary objective:
  To assess whether fear of pain, fear-avoidance beliefs, pain catastrophizing, and sensation seeking as personality traits can explain variations in the present dissociation of sensory-discriminative and emotional-motivational pain responses in chronic pain patients
  Interventions: Behavioral: psychophysical tasks
- Substudy 3 (Experimental): All participants will perform a psychophysical task to assess metacognition in pain perception as an indicator of the cognitive-evaluative pain component. No arms will perform.
  Primary objective:
  To assess whether metacognition on pain perception are involved and subjective ratings of perceived pain and how metacognition relates to pain intensity.
  Secondary objective:
  To assess whether confidentiality as a personality trait , pain catastrophizing, and skin conductance responses are related to metacognition in pain.
  Interventions: Behavioral: cognitive task

INTERVENTIONS:
Behavioral: psychophysical tasks — All participants perform two psychophysical tasks to assess sensory-discriminative and emotional-motivational pain responses independently from each other.
  In addition, in Substudy 1 an operant learning paradigm will be implement to dissociate these responses, increasing the sensory-discriminative pain responses compared to emotional-motivational pain responses by contingent monetary reinforcement or vice versa.
  In Substudy 2, responses of chronic pain patients will be compared to those of healthy participants to characterize possible alterations and operant learning will be operationalized to decrease emotional-motivational pain responses, which are assumed to be already increased in the patients.
  Arms: Substudy 1; Substudy 2
Behavioral: cognitive task — In Substudy 3 participants will perform a psychophysical task to assess metacognition in pain perception as an indicator of the cognitive-evaluative pain component.
  Arms: Substudy 3

SUMMARY:
The experience of pain is more than the conscious perception of nociceptive signals. Emotional and motivational aspects accompany pain, leading to its aversiveness and motivation for avoidance. In chronic pain, a negative hedonic shift has been proposed that is characterized by disproportionally increased emotional-motivational compared to sensory-discriminative pain responses. Such a negative hedonic shift is, for example, mirrored in very high comorbidity rates of chronic pain and affective disorders such as depression and anxiety. The aim of this study is to develop methods that allow the differentiation of sensory-discriminative and emotional-motivational pain response and to characterize mechanisms of the negative hedonic shift.

DETAILED DESCRIPTION:
The experience of pain is more than the conscious perception of nociceptive signals. Emotional and motivational aspects accompany pain, leading to its aversiveness and motivation for avoidance. In chronic pain, a negative hedonic shift has been proposed that is characterized by disproportionally increased emotional-motivational compared to sensory-discriminative pain responses. Such a negative hedonic shift is, for example, mirrored in very high comorbidity rates of chronic pain and affective disorders such as depression and anxiety. However, appropriate psychophysical methods to differentiate sensory-discriminative and emotional-motivational pain processing in humans are lacking. Therefore, only indirect evidence on the assumed negative hedonic shift in chronic pain is available, albeit understanding the mechanisms of such a shift would increase our knowledge on the development and maintenance of chronic pain in important ways with impact beyond pain research. The aim of this study is to develop methods that allow the differentiation of sensory-discriminative and emotional-motivational pain response and to characterize mechanisms of the negative hedonic shift.

A potential benefit of the study will be an increase in the knowledge on mechanisms of the development and maintenance of chronic pain with a focus on emotional-motivational processes likely also relevant in other diseases such as affective disorders.

This study involves only minimal risks for participants. The methods that will be used in the experimental investigations are within the range of standard procedures in pain research and experimental psychology and are frequently used in healthy participants and patients. Experimental pain stimulation will be adjusted to individual pain sensitivity, rendering the applied stimulation tolerable.

Substudy 1 Each participant will perform one testing session of approximately 1.5h duration at the Balgrist Campus, Balgrist University Hospital, Zurich. Healthy volunteers (N=31) will be recruited. The testing session will comprise a discrimination task and an avoidance task to assess sensory-discriminative and emotional-motivational pain components independently of each other. The tasks will be performed in counterbalanced order. After obtaining written informed consent, participants' individual heat pain threshold and tolerance will be determined, based on which the stimulation intensity to be used in the discrimination and the avoidance task will be calculated. After this assessment, participants either perform the discrimination or the avoidance task. Within the discrimination task, participants have to indicate whether they perceived a small increase in temperature or not. In the avoidance task, participants can avoid a painful stimulation by reacting fast enough to a visual cue. Participants will be randomly (balanced randomization) assigned to one of two learning conditions, either reinforcing successful discrimination or avoidance, to increase sensory-discriminative or emotional-motivational pain responses. Reinforcement, implemented by small monetary wins, will start depending on the condition after half the trials of the discrimination or the avoidance task. Subjective ratings of perceived pain intensity and unpleasantness will be assessed within both tasks as control variables to test whether increases in sensory-discriminative or emotional-motivational pain processing generalize to the subjective response channel. At the end of the testing session, participants will complete several questionnaires to investigate whether certain personality traits are related to learning capacity as tested in these tasks.

Substudy 2 Each participant will perform one testing session of approximately 1.5h duration at the Balgrist Campus, Balgrist University Hospital, Zurich. The sample will consist of patients with unspecific musculoskeletal chronic pain (N=31) and age- and sex-matched healthy controls (N=31). As in Substudy 1, the testing session will comprise the discrimination task and the avoidance task to assess sensory-discriminative and emotional-motivational pain components independently of each other. The tasks will be performed in counterbalanced order. After obtaining written informed consent, participants' individual heat pain threshold and tolerance will be determined, based on which the stimulation intensity to be used in the discrimination and the avoidance task will be calculated. After this assessment, participants either perform the discrimination or the avoidance task as in Substudy 1. In contrast to Substudy 1, reinforcement in the avoidance task will be implemented to decrease emotional-motivational pain responses because it is assumed that patients show already increased emotional-motivational compared to sensory-discriminative pain processing. Subjective ratings of perceived pain intensity and unpleasantness will be assessed within both tasks as control variables to test whether increases in sensory-discriminative or emotional-motivational pain processing generalize to the subjective response channel. At the end of the testing session, participants will complete several questionnaires, to investigate whether certain personality traits are related to heightened emotional-motivational pain processing.

Sample sizes for Substudy 1 and 2 are based on a priori sample size calculations using G*Power 3.1 with a desired medium effect size f=0.25, alpha=0.05, beta=0.80, repeated measures ANOVA between-within-subject designs, and an attrition rate of 10%. Outcome variables () will be analyzed in separate mixed model analyses for ANOVA designs with appropriate within- and between-subject factors. Associations of primary endpoints () with personality traits (secondary outcomes) will be analyzed using Person- or Spearman correlation coeffients, where appropriate. Significance levels will be set to 5%, adjusted with false discovery rate for multiple testing. Effect sizes will be calculated in terms of generalized η2 and Cohen's d.

Substudy 3 Each participant will perform one testing session of approximately 1.25h duration at the Balgrist Campus, Balgrist University Hospital, Zurich. Healthy volunteers (N=30) will be recruited. During testing session participants will perform a psychophysical task to assess metacognition in pain perception as an indicator of the cognitive-evaluative pain component. The objective is to assess whether metacognition on pain perception are involved and subjective ratings of perceived pain and how metacognition relates to pain intensity. After obtaining written informed consent, participants' individual heat pain threshold and tolerance will be determined, based on which the stimulation intensity to be used in the experiment will be calculated. After this assessment, participants perform the cognitive pain task. Within this task, participants have to indicate whether they perceived a first or second heat pain stimulus as higher in intensity, whether the higher one was perceived as painful or not, and their confidence in both these answers. In addition, participants will complete several questionnaires to investigate whether certain personality traits and personal states are related to metacognition in pain.

The sample size of Substudy 3 is determined according to Kreft and Leeuw (2007) after which a great enough power will be reached with a sample size of 30 participants and 30 observations to identify cross-level interactions. Substudy 3 follows a within subject design with repeated measures. The tasks that will be performed by each participant include the within-subject factor 'temperature difference' (differences in temperature between first and second stimulus) and the within-subject factor 'temperature level' (temperature relative to individual pain threshold of each stimulus). The order of the different conditions in each task will be applied using a balanced pseudo-randomized order. For testing hypothesis 1ai, 1bi and 1c t-test will be conducted. For Hypothesis 1aii and 1bii chi square tests are planned. To test hypothesis 2a, 2c and 3 logistic hierarchic liner models and for hypothesis 2b and 2d hierarchic linear models will be performed.

Within this study methods that allow the separation of different components of the perception of pain will be developed and validated and which are currently not available. In addition, based on theses methods, a human model on how such components of pain can dissociate will be developed, thereby allowing investigating a prominent assumption on factors that crucially contribute to the development and maintenance of chronic pain. The expected results will form the basis for the development of novel mechanism-based pain therapies.

Psychophysical methods based on experimental psychology and pain research will be used, which have been shown before to be successful in investigating different aspects of pain perception and the modulation of pain perception. The methods used are in the standard range of methods from human pain research and experimental psychology and hold only minimal risk for participants (see above "Risk / Benefit Assessment").

ELIGIBILITY:
For Healthy participants

Inclusion Criteria:

* good overall health status
* sufficient knowledge of German or English to follow instructions
* ability to give written informed consent

Exclusion Criteria:

* pain longer than >3 consecutive days and on more than 30 days within the last 12 months
* major psychiatric or neurological disorders, and substance abuse
* consumption of alcohol, illegal drugs, and analgesic drug within 24 hours before testing

For chronic pain patients

Inclusion Criteria:

* unspecific musculoskeletal chronic pain
* sufficient knowledge of German or English to follow instructions
* ability to give written informed consent

Exclusion Criteria:

* major psychiatric or neurological disorders, excluding depression and anxiety, and substance abuse
* consumption of alcohol, illegal drugs, and analgesic drugs within 24 hours before testing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
ratio of sensory to emotional pain responses | during the procedure
  Ratio of the number of correct responses (%) in a task assessing sensory-discriminative pain responses to number of correct responses (%) in a task assessing emotional-motivational pain responses.

SECONDARY OUTCOMES:
reaction time (RT) | during the procedure
  reaction times
pain threshold | baseline
  Individual pain threshold assessed with experimental heat pain
pain tolerance | baseline
  Individual pain tolerance assessed with experimental heat pain
perceived pain intensity | during the procedure
  Individual perceived pain intensity assessed with experimental heat pain
perceived pain unpleasantness | during the procedure
  Individual perceived pain unpleasantness assessed with experimental heat pain
Fear of Pain Questionnaire (FPQ-III) | during the procedure at day one
  FPQ-III is one questionnaire which is a widely used to assess the fear of pain (FOP) in clinical and non clinical samples. It is one self-report instrument that was developed specifically to assess fear of different stimuli usually causing pain.
  Time duration <5minutes Five point Likert scale Score range (30-150) A higher score indicates higher fear of pain, no cut-off values
Pain Catastrophizing Scale (PCS) | during the procedure at day one
  The PCS was developed in 1995 at the University Centre for Research on Pain and Disability in order to facilitate research on the mechanisms by which catastrophizing impacts on pain experience. Catastrophizing is currently defined as: an exaggerated negative mental set brought to bear during actual or anticipated painful experience.
  Time duration less than 5minutes Five point Likert scale Score range (0-52) <20 low risk for development of chronicity 20-30 moderate risk for development of chronicity >30 high risk for development of chronicity
Fear of Avoidance Beliefs FABQ | during the procedure at day one
  FABQ focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability
  Time duration 5-10minutes Seven point Likert scale Score range (0-96) Higher score indicates fear avoidance behaviors
Personal Evaluation Inventory (PEI) | during procedure
  PEI asses among other things ones trait confidence which might be related to metacognition in pain.
skin conductance responses | during procedure
  individual skin conductance reaction on heat stimuli during the behavioural task
confidence ratings on forced choice questions | during procedure
  Answers on forced-choice questions on which one of two heat stimuli was more intense and whether this one was perceived as painful, ratings of confidence. The answers on the forces-choice questions together with their ratings of confindence in these answers provide a measurement of metacognition.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Becker, PD Dr., Principal Investigator — Balgrist Universitätsklinik
Locations (1):
- Balgrist Campus, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No